CLINICAL TRIAL: NCT03942406
Title: Phase 2b Study of BPZE1 Intranasal Pertussis Vaccine in Adults to Assess Immunological Response and Safety Profile of 1-Dose (Prime) and 2-Doses (Prime+Boost) Schedule, Compared to a Boostrix™ Prime Dose With or Without a BPZE1 Boost Dose
Brief Title: Study of BPZE1 Intranasal Pertussis Vaccine (Administered Via VaxINator(TM)), Prime + Boost, in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ILiAD Biotechnologies (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IB-200P
Record Dates: First submitted 2019-05-02; First posted 2019-05-08 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-05

CONDITIONS: Pertussis; Whooping Cough
Keywords: pertussis; Bordetella infection; Gram-negative bacterial infection; Respiratory tract infection; Whooping cough; Infection; Respiratory tract disease; Vaccine; Immunological factors; Physiological effects of drugs
MeSH Terms: conditions — Whooping Cough; Bordetella Infections; Gram-Negative Bacterial Infections; Respiratory Tract Infections; Infections; Respiratory Tract Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- BPZE1 Intranasal Prime, BPZE1 Boost (Experimental): Individual will receive an intranasal dose of BPZE1 via the VaxINator atomization device and a dose of intramuscular (I.M.) placebo. Individuals will receive a boost dose of intranasal BPZE1 via the VaxINator™ atomization device.
  Interventions: Combination Product: BPZE1 pertussis vaccine and VaxINator(TM) Atomization Device
- BPZE1 Intranasal Prime, Placebo Boost (Experimental): Individual will receive an intranasal dose of BPZE1 via the VaxINator atomization device and a dose of intramuscular (I.M.) placebo. Individuals will receive a boost dose of intranasal placebo via the VaxINator™ atomization device.
  Interventions: Combination Product: BPZE1 pertussis vaccine and VaxINator(TM) Atomization Device
- Boostrix IM Prime, BPZE1 Boost (Experimental): Individual will receive an intranasal dose of placebo via the VaxINator atomization device and a dose of intramuscular (I.M.) Boostrix (aP vaccine comparator). Individuals will receive a boost dose of intranasal BPZE1 via the VaxINator™ atomization device.
  Interventions: Combination Product: BPZE1 pertussis vaccine and VaxINator(TM) Atomization Device
- Boostrix IM Prime, Placebo Boost (Active Comparator): Individual will receive an intranasal dose of placebo via the VaxINator atomization device and a dose of intramuscular (I.M.) Boostrix (aP vaccine comparator). Individuals will receive a boost dose of intranasal placebo via the VaxINator™ atomization device.
  Interventions: Combination Product: BPZE1 pertussis vaccine and VaxINator(TM) Atomization Device

INTERVENTIONS:
Combination Product: BPZE1 pertussis vaccine and VaxINator(TM) Atomization Device — Live attenuated pertussis vaccine administered via the VaxINator(TM) atomization device

SUMMARY:
This study evaluates the safety and immunogenicity of the BPZE1 live attenuated pertussis vaccine, intended to prevent nasopharyngeal colonization and pertussis disease, and compares a single (prime) BPZE1 dose or BPZE1 2-dose (prime + boost) to a single (prime) Boostrix or Boostrix prime + BPZE1 boost.

DETAILED DESCRIPTION:
This study evaluates the safety and immunogenicity of the BPZE1 live attenuated pertussis vaccine, intended to prevent nasopharyngeal colonization and pertussis disease, and compares a single (prime) BPZE1 dose or BPZE1 2-dose (prime + boost) to a single (prime) Boostrix or Boostrix prime + BPZE1 boost. This is a multi-center, randomized, placebo-controlled, and observer blinded trial in healthy adults with a 6 month safety follow-up after the last vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Is a male or nonpregnant female 18 to 50 years of age, inclusive, on Day 1 (primary vaccination).
2. Is capable of understanding the written informed consent, provides signed and witnessed written informed consent, and agrees to comply with protocol requirements.
3. Female subjects must be nonpregnant and nonlactating and meet 1 of the following criteria:

   1. Postmenopausal (defined as 12 consecutive months with no menses without an alternative medical cause or documented plasma follicle-stimulating hormone level in the postmenopausal range);
   2. Surgically sterile (ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy).

      NOTE: These procedures and laboratory test results must be confirmed by physical examination, or by subject recall of specific date and hospital/facility of procedure, or by medical documentation of said procedure.
   3. Is of childbearing potential (defined as any female who has experienced menarche and who is NOT permanently sterile or postmenopausal), agrees to be heterosexually inactive from at least 21 days prior to enrollment and through 3 months after the boosting vaccination or agrees to consistently use any of the following methods of contraception from at least 21 days prior to enrollment and through 3 months after the boosting vaccination:

   i. Condoms (male or female) with spermicide ii. Diaphragm with spermicide iii. Cervical cap with spermicide iv. Intrauterine device v. Oral or patch contraceptives vi. Norplant®, Depo-Provera®, or other FDA approved contraceptive method that is designed to protect against pregnancy.

   NOTE: Periodic abstinence (eg, calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are not acceptable methods of contraception.
4. Has a stable health status as assessed by the investigator, as established by physical examination, vital sign measurements, and medical history.
5. Has access to a consistent and reliable means of telephone contact, which may be in the home, workplace, or by personal mobile electronic device.
6. Is able to understand and comply with planned study procedures.
7. Lives a reasonable distance from the clinical site to be able to travel to and from the clinical site for follow-up visits and agrees to go to the clinical site for evaluation (or provide medical record access if evaluated elsewhere) in the event of an AE.
8. Agrees to stay in contact with the clinical site for the duration of the study, has no current plans to move from the study area, and provides updated contact information as necessary.

Exclusion Criteria:

1. History of being vaccinated in the past 5 years against pertussis.
2. Any significant past reaction to any component of Boostrix (at the discretion of the investigator).
3. Subject reported diagnosis of pertussis in the past 10 years (must be laboratory confirmed or physician diagnosed from medical records).
4. Vital signs by FDA toxicity scoring >1 (may be repeated once during the screening period to allow for inclusion and the most recent measurement taken at baseline).
5. Chronic illness being treated actively and with evidence of recent intervention for worsening or fluctuating symptoms (at the discretion of the investigator).
6. The subject has a history of active cancer (malignancy) in the last 10 years (exception is subjects with adequately treated non melanomatous skin carcinoma, who may participate in the study).
7. Current use of any smoking products and unwillingness to refrain from the use of any smoking products from screening through 28 days after the boosting vaccination.
8. Use of narcotic drugs, evidenced by urine toxicology screen or a history of drug/alcohol abuse within the past 2 years.
9. Has donated blood or suffered from blood loss of more than 450 mL (1 unit of blood) within 60 days prior to screening or donated plasma within 14 days prior to screening.
10. Receipt of immunoglobulin, blood-derived products, systemic corticosteroids, or other immunosuppressant drugs within 90 days prior to Day 1.
11. Asthma, obstructive nasal canal, recurrent or acute sinusitis or other chronic respiratory problems inclusive of the diagnosis of any significant pulmonary disease.
12. History of nasal surgery or Bell's palsy.
13. Use of repeated nasal sprays, Neti pot, routine nasal washing within the past 1 month (more than 2 times per week). Subjects must agree to refrain from use of any of these modalities through Day 113.
14. A temporary exclusion to vaccinate if acute respiratory tract infection or rhinorrhea or temperature >100.4°F (no symptoms for 3 days prior to vaccination day). Subjects may be vaccinated if they stay within the vaccination window (screening [30 days] or at the time of the booster [10 days]).

    NOTE: If a subject exceeds the screening window, they must be reconsented and screening must be reinitiated.
15. Use of corticosteroids in the respiratory tract (eg, nasal steroids, inhaled steroids) within 30 days prior to Day 1.
16. Receipt of a licensed vaccine within the last 30 days prior to Day 1 or planned vaccination during the active study conduct through Day 113. In the case of seasonal influenza, vaccination should not be withheld and is not contraindicated for subject participation. However, vaccination should be planned outside of a 30 day pre- and 30 day post vaccination window whenever possible.
17. Known hypersensitivity to any component of the study vaccines.
18. Participation in any other clinical trial for the testing of an unlicensed product during the previous 6 months or planned during the study conduct.
19. Inability to adhere to the protocol, including plans to move from the area.
20. Personal history or family (first degree) history of congenital or hereditary immunodeficiency.
21. Past or present infection with human immunodeficiency virus, hepatitis B, or hepatitis C by screening test.
22. Any autoimmune or immunodeficiency disease/condition (inherited or iatrogenic).
23. Any neurological disease or history of significant neurological disorder (eg, meningitis, seizures, multiple sclerosis, vasculitis, migraines, Guillain-Barré syndrome [genetic/congenital or acquired]).
24. Any medical condition that, in the opinion of the investigator, might interfere with the evaluation of the study objectives or might affect the safety of the individual, (eg, major depression or history of suicidal attempt).
25. Toxicity grading >1 for screening laboratory test results for kidney, hepatic, and hematologic values (may be repeated once during the screening period to allow for inclusion and the most recent measurement taken at baseline). See Table 13 2 for specifically designated parameters.
26. Body mass index <17 kg/m2 or >40 kg/m2.
27. Frequent contact with children less than 1 year of age (parent, childcare worker, nurse, etc.) or residence in the same household as persons with known immunodeficiency including persons on immunosuppressant therapy.
28. Study team member or first-degree relative of study team member.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary B Manning, MD, Principal Investigator — Rapid Medical Research Inc; Barbara Rizzardi, MD, Principal Investigator — Advanced Clinical Research Services, LLC; Vicki Miller, MD, Principal Investigator — DM Clinical Research
Locations (3):
- United States (3):
  - Rapid medical Research Inc, Cleveland, Ohio
  - DM Clinical Research, Tomball, Texas
  - Advanced Clinical Research, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Althouse BM, Scarpino SV. Asymptomatic transmission and the resurgence of Bordetella pertussis. BMC Med. 2015 Jun 24;13:146. doi: 10.1186/s12916-015-0382-8. PMID 26103968
- [Background] Feunou PF, Ismaili J, Debrie AS, Huot L, Hot D, Raze D, Lemoine Y, Locht C. Genetic stability of the live attenuated Bordetella pertussis vaccine candidate BPZE1. Vaccine. 2008 Oct 23;26(45):5722-7. doi: 10.1016/j.vaccine.2008.08.018. Epub 2008 Aug 30. PMID 18762220
- [Background] Feunou PF, Mielcarek N, Locht C. Reciprocal interference of maternal and infant immunization in protection against pertussis. Vaccine. 2016 Feb 17;34(8):1062-9. doi: 10.1016/j.vaccine.2016.01.011. Epub 2016 Jan 15. PMID 26776471
- [Background] Locht C, Papin JF, Lecher S, Debrie AS, Thalen M, Solovay K, Rubin K, Mielcarek N. Live Attenuated Pertussis Vaccine BPZE1 Protects Baboons Against Bordetella pertussis Disease and Infection. J Infect Dis. 2017 Jul 1;216(1):117-124. doi: 10.1093/infdis/jix254. PMID 28535276
- [Background] Mielcarek N, Debrie AS, Raze D, Bertout J, Rouanet C, Younes AB, Creusy C, Engle J, Goldman WE, Locht C. Live attenuated B. pertussis as a single-dose nasal vaccine against whooping cough. PLoS Pathog. 2006 Jul;2(7):e65. doi: 10.1371/journal.ppat.0020065. PMID 16839199
- [Background] Mielcarek N, Debrie AS, Mahieux S, Locht C. Dose response of attenuated Bordetella pertussis BPZE1-induced protection in mice. Clin Vaccine Immunol. 2010 Mar;17(3):317-24. doi: 10.1128/CVI.00322-09. Epub 2010 Jan 27. PMID 20107007
- [Background] Skerry CM, Cassidy JP, English K, Feunou-Feunou P, Locht C, Mahon BP. A live attenuated Bordetella pertussis candidate vaccine does not cause disseminating infection in gamma interferon receptor knockout mice. Clin Vaccine Immunol. 2009 Sep;16(9):1344-51. doi: 10.1128/CVI.00082-09. Epub 2009 Jul 22. PMID 19625486
- [Background] Warfel JM, Zimmerman LI, Merkel TJ. Acellular pertussis vaccines protect against disease but fail to prevent infection and transmission in a nonhuman primate model. Proc Natl Acad Sci U S A. 2014 Jan 14;111(2):787-92. doi: 10.1073/pnas.1314688110. Epub 2013 Nov 25. PMID 24277828
- [Derived] Keech C, Miller VE, Rizzardi B, Hoyle C, Pryor MJ, Ferrand J, Solovay K, Thalen M, Noviello S, Goldstein P, Gorringe A, Cavell B, He Q, Barkoff AM, Rubin K, Locht C. Immunogenicity and safety of BPZE1, an intranasal live attenuated pertussis vaccine, versus tetanus-diphtheria-acellular pertussis vaccine: a randomised, double-blind, phase 2b trial. Lancet. 2023 Mar 11;401(10379):843-855. doi: 10.1016/S0140-6736(22)02644-7. PMID 36906345
- See also: DHHS, FDA, CBER (US). Guidance for industry: Toxicity grading for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials — http://www.gpo.gov/fdsys/pkg/FR-2007-09-27/pdf/E7-19155.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Period 1 (Day 1): Prime; Period 2 (Day 85): Boost
  300 participants:
  * 20 received BPZE1 10^7 CFU as a Safety Lead-in cohort (Prime/Boost: BPZE1/BPZE1 [n=8]; BPZE1/Placebo [n=8]; Boostrix/BPZE1 [n=4]). Safety Lead-in cohort used for one secondary endpoint (abnormal laboratory) and Safety.
  * 280 in 10^9 ITT Analysis Set (Prime/Boost: BPZE 10^9/BPZE1 10^9 [n=92]; BPZE1 10^9/Placebo [n=92]; Boostrix/BPZE1 10^9 [n=46], and Boostrix/Placebo [n=50]).
Groups:
- BPZE1 Intranasal Prime, BPZE1 Boost: Individual will receive an intranasal dose of BPZE1 via the VaxINator atomization device and a dose of intramuscular (IM) placebo on Day 1. Individuals will receive a boost dose of intranasal BPZE1 via the VaxINator™ atomization device on Day 85.
  (10^9 ITT Analysis Set)
- BPZE1 Intranasal Prime, Placebo Boost: Individual will receive an intranasal dose of BPZE1 via the VaxINator atomization device and a dose of IM placebo on Day 1. Individuals will receive a boost dose of intranasal placebo via the VaxINator™ atomization device on Day 85.
  (10^9 ITT Analysis Set)
- Boostrix IM Prime, BPZE1 Boost: Individual will receive an intranasal dose of placebo via the VaxINator atomization device and a dose of IM Boostrix (aP vaccine comparator) on Day 1. Individuals will receive a boost dose of intranasal BPZE1 via the VaxINator™ atomization device on Day 85.
  (10^9 ITT Analysis Set)
- Boostrix IM Prime, Placebo Boost: Individual will receive an intranasal dose of placebo via the VaxINator atomization device and a dose of IM Boostrix (aP vaccine comparator) on Day 1. Individuals will receive a boost dose of intranasal placebo via the VaxINator™ atomization device on Day 85.
  (10^9 ITT Analysis Set)
- BPZE1 (10^7) Intranasal Prime, BPZE1 (10^7) Boost: Individual will receive an intranasal dose of BPZE1 via the VaxINator atomization device and a dose of IM placebo on Day 1. Individuals will receive a boost dose of intranasal BPZE1 via the VaxINator™ atomization device on Day 85.
  (10^7 Safety Lead-in Analysis Set)
- BPZE1 (10^7) Intranasal Prime, Placebo Boost: Individual will receive an intranasal dose of BPZE1 via the VaxINator atomization device and a dose of IM placebo on Day 1. Individuals will receive a boost dose of intranasal placebo via the VaxINator™ atomization device on Day 85.
  (10^7 Safety Lead-in Analysis Set)
- Boostrix IM Prime, BPZE1 (10^7) Boost: Individual will receive an intranasal dose of placebo via the VaxINator atomization device and a dose of IM Boostrix (aP vaccine comparator) on Day 1. Individuals will receive a boost dose of intranasal BPZE1 via the VaxINator™ atomization device on Day 85.
  (10^7 Safety Lead-in Analysis Set)
Period: Overall Study
Arm/Group | BPZE1 Intranasal Prime, BPZE1 Boost | BPZE1 Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 Boost | Boostrix IM Prime, Placebo Boost | BPZE1 (10^7) Intranasal Prime, BPZE1 (10^7) Boost | BPZE1 (10^7) Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 (10^7) Boost
Started | 92 | 92 | 46 | 50 | 8 | 8 | 4
Completed | 81 | 85 | 41 | 40 | 6 | 7 | 4
Not Completed | 11 | 7 | 5 | 10 | 2 | 1 | 0
Not completed — Lost to Follow-up | 4 | 5 | 3 | 7 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 3 | 0 | 0 | 0
Not completed — Other: early termination, telemedicine visits | 4 | 1 | 1 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- BPZE1 Intranasal Prime, BPZE1 Boost: Individual will receive an intranasal dose of BPZE1 via the VaxINator atomization device and a dose of IM placebo on Day. Individuals will receive a boost dose of intranasal BPZE1 via the VaxINator™ atomization device on Day 85.
  (10^9 ITT Analysis Set)
- Total: Total of all reporting groups
Arm/Group | BPZE1 Intranasal Prime, BPZE1 Boost | BPZE1 Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 Boost | Boostrix IM Prime, Placebo Boost | BPZE1 (10^7) Intranasal Prime, BPZE1 (10^7) Boost | BPZE1 (10^7) Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 (10^7) Boost | Total
Number analyzed (Participants) | 92 | 92 | 46 | 50 | 8 | 8 | 4 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (9.0) | 35.2 (8.8) | 34.6 (9.0) | 34.2 (9.9) | 31.6 (10.3) | 34.6 (8.7) | 35.5 (12.0) | 35.0 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 46 | 26 | 27 | 3 | 4 | 3 | 165
  Male | 36 | 46 | 20 | 23 | 5 | 4 | 1 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 11 | 8 | 7 | 0 | 1 | 0 | 42
  Not Hispanic or Latino | 77 | 81 | 38 | 43 | 8 | 7 | 4 | 258
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 5 | 1 | 0 | 0 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 3
  Black or African American | 19 | 22 | 9 | 8 | 0 | 1 | 2 | 61
  White | 70 | 65 | 31 | 41 | 7 | 7 | 2 | 223
  More than one race | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 4
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.0 (5.4) | 28.1 (5.6) | 27.7 (5.0) | 27.2 (5.0) | 26.7 (7.7) | 31.1 (7.0) | 29.6 (7.3) | 27.9 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Nasal Mucosal Seroconversion (Immunoglobulin A [IgA])
Description: Number of participants who achieve mucosal seroconversion (IgA) against at least 1 anti-pertussis antibody for whole cell extract (WCE), pertussis toxin (PT), filamentous hemagglutinin (FHA), or pertactin (PRN) on Day 29 or Day 113. Mucosal seroconversion was defined as a 2-fold increase over the baseline value or a 4-fold increase over the minimal detection limit of the assay (whenever the baseline value was below the detection limits of the assay).
Time Frame: Days 29 and 113
Population: 10^9 Immunogenicity Analysis Set. The overall number of participants analyzed includes participants with nonmissing values. Note: Participants who were randomized to receive BPZE1 as the second vaccination (ie, revaccination/attenuated challenge) but who did not receive a second vaccination and continued in the study after second vaccination were placed into the BPZE1/Placebo or Boostrix/Placebo group according to first vaccine received.
Measure: Count of Participants; unit: Participants
Groups:
- BPZE1 Intranasal Prime, BPZE1 Boost: Individual will receive an intranasal dose of BPZE1 via the VaxINator atomization device and a dose of IM placebo on Day 1. Individuals will receive a boost dose of intranasal BPZE1 via the VaxINator™ atomization device on Day 85.
- BPZE1 Intranasal Prime, Placebo Boost: Individual will receive an intranasal dose of BPZE1 via the VaxINator atomization device and a dose of IM placebo on Day 1. Individuals will receive a boost dose of intranasal placebo via the VaxINator™ atomization device on Day 85.
- Boostrix IM Prime, BPZE1 Boost: Individual will receive an intranasal dose of placebo via the VaxINator atomization device and a dose of IM Boostrix (aP vaccine comparator) on Day 1. Individuals will receive a boost dose of intranasal BPZE1 via the VaxINator™ atomization device on Day 85.
- Boostrix IM Prime, Placebo Boost: Individual will receive an intranasal dose of placebo via the VaxINator atomization device and a dose of IM Boostrix (aP vaccine comparator) on Day 1. Individuals will receive a boost dose of intranasal placebo via the VaxINator™ atomization device on Day 85.
Arm/Group | BPZE1 Intranasal Prime, BPZE1 Boost | BPZE1 Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 Boost | Boostrix IM Prime, Placebo Boost
Number analyzed (Participants) | 84 | 94 | 42 | 45
Participants | 79 | 89 | 38 | 42

2. Primary Outcome: Safety - Number of Participants With Nasal/Respiratory Solicited Adverse Events (AEs)
Description: Number of participants with Solicited AEs (nasal/respiratory reactogenicity events) by Grade - Any Day Grade 1 through 3 and Grade 3. Grading of reactogenicity is defined per protocol as Grade 1 (mild), Grade 2 (moderate), and Grade 3 (severe) AEs.
Time Frame: Through 7 Days Following Day 1 Vaccination
Population: 10^9 Safety Analysis Set. Note: Participants who were randomized to receive BPZE1 as the second vaccination (ie, revaccination/attenuated challenge) but who did not receive a second vaccination and continued in the study were placed into the BPZE1/Placebo or Boostrix/Placebo group according to first vaccine received.
Measure: Number; unit: participants
Arm/Group | BPZE1 Intranasal Prime, BPZE1 Boost | BPZE1 Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 Boost | Boostrix IM Prime, Placebo Boost
Number analyzed (Participants) | 87 | 96 | 46 | 50
participants
  Runny Nose - Any Day Grade 1 through 3 | 25 | 41 | 17 | 16
  Runny Nose - Any Day Grade 3 | 0 | 0 | 0 | 0
  Stuffy Nose/Congestion - Any Day Grade 1 through 3 | 27 | 44 | 19 | 15
  Stuffy Nose/Congestion - Any Day Grade 3 | 0 | 0 | 0 | 0
  Nasal Pain/Irritation - Any Day Grade 1 through 3 | 10 | 13 | 7 | 7
  Nasal Pain/Irritation - Any Day Grade 3 | 0 | 0 | 0 | 0
  Epistaxis - Any Day Grade 1 through 3 | 1 | 5 | 2 | 1
  Epistaxis - Any Day Grade 3 | 0 | 0 | 0 | 0
  Sneezing - Any Day Grade 1 through 3 | 25 | 35 | 15 | 13
  Sneezing - Any Day Grade 3 | 0 | 0 | 0 | 0
  Sinus Pressure/Pain - Any Day Grade 1 through 3 | 12 | 19 | 5 | 10
  Sinus Pressure/Pain - Any Day Grade 3 | 0 | 0 | 0 | 0
  Sore/Irritated Throat - Any Day Grade 1 through 3 | 22 | 29 | 8 | 10
  Sore/Irritated Throat - Any Day Grade 3 | 0 | 0 | 0 | 0
  Cough - Any Day Grade 1 through 3 | 11 | 18 | 10 | 9
  Cough - Any Day Grade 3 | 0 | 0 | 0 | 0
  Shortness of Breath/Wheezing - Any Day Grade 1 through 3 | 1 | 7 | 2 | 3
  Shortness of Breath/Wheezing - Any Day Grade 3 | 0 | 0 | 0 | 0

3. Primary Outcome: Safety - Number of Participants With Local Solicited AEs
Description: Number of participants with Solicited AEs (local reactogenicity events) by Grade - Any Day Grade 1 through 4 and Grade 3 and 4. Grading of reactogenicity is defined per protocol as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), and Grade 4 (potentially life-threatening) AEs.
Time Frame: Through 7 Days Following Day 1 Vaccination
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | BPZE1 Intranasal Prime, BPZE1 Boost | BPZE1 Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 Boost | Boostrix IM Prime, Placebo Boost
Number analyzed (Participants) | 87 | 96 | 46 | 50
participants
  Pain - Any Day Grade 1 Through 4 | 8 | 7 | 22 | 27
  Pain - Any Day Grade 3 and 4 | 0 | 0 | 0 | 0
  Tenderness - Any Day Grade 1 Through 4 | 15 | 13 | 28 | 30
  Tenderness - Any Day Grade 3 and 4 | 0 | 0 | 0 | 0
  Erythema/Redness - Any Day Grade 1 Through 4 | 0 | 2 | 1 | 2
  Erythema/Redness - Any Day Grade 3 and 4 | 0 | 0 | 0 | 0
  Induration/Swelling - Any Day Grade 1 Through 4 | 0 | 0 | 4 | 2
  Induration/Swelling - Any Day Grade 3 and 4 | 0 | 0 | 0 | 0

4. Primary Outcome: Safety - Number of Participants With Systemic Solicited AEs
Description: Number of participants with Solicited AEs (systemic reactogenicity events) by Grade - Any Day Grade 1 through 3 and Grade 3. Grading of reactogenicity is defined per protocol as Grade 1 (mild), Grade 2 (moderate), and Grade 3 (severe) AEs.
Time Frame: Through 7 Days Following Day 1 Vaccination
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | BPZE1 Intranasal Prime, BPZE1 Boost | BPZE1 Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 Boost | Boostrix IM Prime, Placebo Boost
Number analyzed (Participants) | 87 | 96 | 46 | 50
participants
  Fever - Any Day Grade 1 through 3 | 0 | 1 | 0 | 0
  Fever - Any Day Grade 3 | 0 | 1 | 0 | 0
  Fatigue (Tiredness) - Any Day Grade 1 through 3 | 27 | 35 | 9 | 12
  Fatigue (Tiredness) - Any Day Grade 3 | 0 | 1 | 0 | 0
  Malaise (General Unwell Feeling) - Any Day Grade 1 through 3 | 13 | 25 | 6 | 8
  Malaise (General Unwell Feeling) - Any Day Grade 3 | 0 | 1 | 0 | 0
  Myalgia (Body Aches/Muscular Pain) - Any Day Grade 1 through 3 | 8 | 19 | 4 | 8
  Myalgia (Body Aches/Muscular Pain) - Any Day Grade 3 | 0 | 1 | 0 | 0
  Arthralgia (Joint Pain) - Any Day Grade 1 through 3 | 5 | 7 | 1 | 4
  Arthralgia (Joint Pain) - Any Day Grade 3 | 0 | 0 | 0 | 0
  Headache - Any Day Grade 1 through 3 | 31 | 37 | 13 | 22
  Headache - Any Day Grade 3 | 0 | 1 | 0 | 0
  Rash/Hypersensitivity - Any Day Grade 1 through 3 | 0 | 4 | 0 | 1
  Rash/Hypersensitivity - Any Day Grade 3 | 0 | 1 | 0 | 0

5. Primary Outcome: Safety Lead-in Participants With Abnormal Laboratory Parameters (BPZE1 10^7 Safety Lead-In)
Description: Number of participants in the safety lead-in cohort with Grade 2 through 4 laboratory abnormalities: Serum Chemistry - Bilirubin, Creatinine, ALT, AST; WBC, Hemoglobin, Prothrombin time, Partial Thromboplastin Time. Grading of laboratory results is defined per protocol as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (potentially life-threatening) laboratory abnormalities (DHHS 2007).
Time Frame: Days 8 and 92
Population: Safety Lead-in Participants vaccinated with BPZE1 10^7 CFU for Prime (Day 1) and/or Boost (Day 85)
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 Intranasal Prime, BPZE1 Boost | BPZE1 Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 Boost
Number analyzed (Participants) | 8 | 8 | 4
Participants
  Bilirubin Increase Day 8 | 1 | 0 | 0
  Bilirubin Increase Day 92 | 0 | 0 | 0
  Creatinine Day 8 | 0 | 0 | 0
  Creatinine Day 92 | 0 | 0 | 0
  ALT Day 8 | 0 | 0 | 0
  ALT Day 92 | 0 | 0 | 0
  AST Day 8 | 0 | 0 | 0
  AST Day 92 | 0 | 0 | 0
  WBC decrease Day 8 | 0 | 0 | 0
  WBC decrease Day 92 | 0 | 0 | 0
  WBC Increase Day 8 | 0 | 0 | 0
  WBC Increase Day 92 | 0 | 0 | 0
  Hemoglobin Day 8 | 0 | 0 | 1
  Hemoglobin Day 92 | 0 | 0 | 1
  Platelets Decrease Day 8 | 0 | 0 | 0
  Platelets Decrease Day 92 | 0 | 0 | 0
  Prothrombin Time Increase by Factor Day 8 | 2 | 0 | 0
  Prothrombin Time Increase by Factor Day 92 | 0 | 0 | 0
  Partial Thromboplastin Time Increase by Factor Day 8 | 0 | 0 | 0
  Partial Thromboplastin Time Increase by Factor Day 92 | 0 | 0 | 0

6. Secondary Outcome: Systemic Immunogenicity - Summary of Systemic IgG Seroconversion Endpoints
Description: Number of participants who achieve seroconversion (serum IgG) against 1 or more pertussis antigens (pertussis toxin [PT], filamentous hemagglutinin [FHA], pertactin [PRN], or whole cell extract [WCE]) on Days 29, 85, 113, 169, and/or 254. Systemic seroconversion was defined as a 2-fold increase over the baseline value or a 4-fold increase over the minimal detection limit of the assay (whenever the baseline value fell below the detection limits of the assay).
Time Frame: 9 months
Population: 10^9 Immunogenicity Analysis Set. The number analyzed includes participants with nonmissing values. Note: Participants who were randomized to receive BPZE1 as the second vaccination (ie, revaccination/attenuated challenge) but who did not receive a second vaccination and continued in the study after second vaccination were placed into the BPZE1/Placebo or Boostrix/Placebo group according to first vaccine received.
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 Intranasal Prime, BPZE1 Boost | BPZE1 Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 Boost | Boostrix IM Prime, Placebo Boost
Number analyzed (Participants) | 85 | 94 | 43 | 45
Participants
  At least 1 of WCE, PT, FHA, PRN: Any of Days 29, 85, or 113 | 63 | 71 | 41 | 45
  At least 1 of WCE, PT, FHA, PRN: Either Day 169 or Day 254: number analyzed (Participants) | 77 | 89 | 38 | 39
  At least 1 of WCE, PT, FHA, PRN: Either Day 169 or Day 254 | 54 | 59 | 33 | 32
  WCE: Either Day 29 or Day 113 | 45 | 41 | 28 | 32
  PT, FHA, PRN: Either Day 29 or Day 113 | 19 | 16 | 28 | 28
  At least 2 of WCE, PT, FHA, OR PRN: Any of Days 29, 85, or 113 | 46 | 50 | 37 | 41
  At least 2 of WCE, PT, FHA, OR PRN: Either Day 169 or Day Day 254: number analyzed (Participants) | 77 | 89 | 38 | 39
  At least 2 of WCE, PT, FHA, OR PRN: Either Day 169 or Day Day 254 | 40 | 41 | 32 | 28
  Boosting Achieved on Day 113 (over Day 85) Against WCE: number analyzed (Participants) | 77 | 87 | 39 | 39
  Boosting Achieved on Day 113 (over Day 85) Against WCE | 8 | 4 | 4 | 2

7. Secondary Outcome: Systemic Immunogenicity - Summary of Systemic IgA Seroconversion Endpoints
Description: Number of participants who achieve seroconversion (serum IgA) against 1 or more pertussis antigens (PT, FHA, PRN) on Days 29, 85, 113, 169, and/or 254. Systemic seroconversion was defined as a 2-fold increase over the baseline value or a 4-fold increase over the minimal detection limit of the assay (whenever the baseline value fell below the detection limits of the assay).
Time Frame: 9 Months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 Intranasal Prime, BPZE1 Boost | BPZE1 Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 Boost | Boostrix IM Prime, Placebo Boost
Number analyzed (Participants) | 85 | 94 | 43 | 45
Participants
  Against at least 1 of PT, FHA, or PRN: Any of Days 29, 85, or 113 | 64 | 71 | 40 | 41
  Against at least 1 of PT, FHA, or PRN: Either day 169 or Day 254: number analyzed (Participants) | 77 | 89 | 38 | 39
  Against at least 1 of PT, FHA, or PRN: Either day 169 or Day 254 | 55 | 58 | 32 | 29
  Against PT, FHA, and PRN: Either Day 29 or Day 113 | 23 | 29 | 18 | 9
  Against at least 2 of PT, FHA, or PRN: Each Day 29, 85, or 113: number analyzed (Participants) | 77 | 86 | 39 | 39
  Against at least 2 of PT, FHA, or PRN: Each Day 29, 85, or 113 | 25 | 28 | 14 | 13
  Against at least 2 of PT, FHA, or PRN: Any of Days 29, 85, or 113 | 50 | 49 | 28 | 30
  Against at least 2 of PT, FHA, or PRN: Either Day 169 or Day 254: number analyzed (Participants) | 77 | 89 | 38 | 39
  Against at least 2 of PT, FHA, or PRN: Either Day 169 or Day 254 | 41 | 30 | 24 | 14
  Boosting Achieved on Day 113 (over Day 85) against PT: number analyzed (Participants) | 77 | 87 | 39 | 39
  Boosting Achieved on Day 113 (over Day 85) against PT | 3 | 2 | 4 | 0
  Boosting Achieved on Day 113 (over Day 85) against FHA: number analyzed (Participants) | 77 | 87 | 39 | 39
  Boosting Achieved on Day 113 (over Day 85) against FHA | 6 | 4 | 3 | 1
  Boosting Achieved on Day 113 (over Day 85) against PRN: number analyzed (Participants) | 77 | 87 | 39 | 39
  Boosting Achieved on Day 113 (over Day 85) against PRN | 13 | 4 | 8 | 0

8. Secondary Outcome: Systemic Immunogenicity - Summary of Geometric Mean Fold Rises (GMFRs) of Systemic IgG Against Whole Cell Extract by Vaccine Group and Time Point
Description: Systemic Immunogenicity: Summary of GMFRs of Systemic IgG Against Whole Cell Extract by Vaccine Group and Time Point - GMFRs on Day 29 and Day 85 over baseline (Day 1)
Time Frame: Days 29 and 85
Population: 10^9 Immunogenicity Analysis Set. The Day 29 and Day 85 GMFR values are for the pooled BPZE1 group (BPZE1/BPZE1 and BPZE1/placebo) and pooled Boostrix group (Boostrix/BPZE1 and Boostrix/placebo), since these Days were prior to the Day 85 challenge/boost. The number analyzed includes participants with nonmissing values.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- BPZE1 Intranasal Prime: Individual will receive an intranasal dose of BPZE1 via the VaxINator atomization device and a dose of IM placebo on Day 1.
- Boostrix IM Prime: Individual will receive an intranasal dose of placebo via the VaxINator atomization device and a dose of IM Boostrix (aP vaccine comparator) on Day 1.
Arm/Group | BPZE1 Intranasal Prime | Boostrix IM Prime
Number analyzed (Participants) | 179 | 88
Ratio
  GMFR WCE Day 29: number analyzed (Participants) | 178 | 88
  GMFR WCE Day 29 | 1.80 [1.63 to 2.00] | 3.06 [2.57 to 3.64]
  GMFR WCE Day 85: number analyzed (Participants) | 172 | 82
  GMFR WCE Day 85 | 1.76 [1.59 to 1.94] | 2.30 [1.94 to 2.72]

9. Secondary Outcome: Systemic Immunogenicity - Summary of GMFRs of Systemic IgG Against Whole Cell Extract by Vaccine Group and Time Point
Description: Systemic Immunogenicity: Summary of GMFRs of Systemic IgG Against Whole Cell Extract by Vaccine Group and Time Point - GMFRs on Days 113, 169, and 254 over baseline (Day 1)
Time Frame: Days 113, 169 and 254
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | BPZE1 Intranasal Prime, BPZE1 Boost | BPZE1 Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 Boost | Boostrix IM Prime, Placebo Boost
Number analyzed (Participants) | 85 | 94 | 43 | 45
Ratio
  GMFR WCE Day 113: number analyzed (Participants) | 77 | 89 | 43 | 45
  GMFR WCE Day 113 | 2.10 [1.79 to 2.48] | 1.64 [1.42 to 1.89] | 2.73 [2.01 to 3.71] | 2.04 [1.63 to 2.56]
  GMFR WCE Day 169: number analyzed (Participants) | 76 | 86 | 37 | 39
  GMFR WCE Day 169 | 1.85 [1.57 to 2.18] | 1.54 [1.34 to 1.78] | 2.32 [1.67 to 3.22] | 1.62 [1.33 to 1.98]
  GMFR WCE Day 254: number analyzed (Participants) | 73 | 85 | 37 | 37
  GMFR WCE Day 254 | 1.66 [1.41 to 1.96] | 1.43 [1.26 to 1.61] | 1.99 [1.52 to 2.59] | 1.37 [1.12 to 1.66]

10. Secondary Outcome: Mucosal Immunogenicity - Summary of Mucosal Absolute S-IgA/Total S-IgA Seroconversion Endpoints
Description: Number of participants who achieve seroconversion against any pertussis specific antigen (PT, PRN, FHA, or WCE) in nasal secretions (S-IgA). Mucosal seroconversion was defined as a 2-fold increase over the baseline value or a 4-fold increase over the minimal detection limit of the assay (whenever the baseline value was below the detection limits of the assay).
Time Frame: 9 months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 Intranasal Prime, BPZE1 Boost | BPZE1 Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 Boost | Boostrix IM Prime, Placebo Boost
Number analyzed (Participants) | 85 | 94 | 43 | 45
Participants
  Against at least 1 of WCE, PT, FHA, or PRN: Any of Days 29, 78, or 113: number analyzed (Participants) | 83 | 94 | 42 | 45
  Against at least 1 of WCE, PT, FHA, or PRN: Any of Days 29, 78, or 113 | 75 | 84 | 33 | 27
  Against at least 1 of WCE, PT, FHA, or PRN: Either Day 169 or Day 254: number analyzed (Participants) | 75 | 90 | 37 | 39
  Against at least 1 of WCE, PT, FHA, or PRN: Either Day 169 or Day 254 | 66 | 63 | 30 | 13
  Against WCE: Either Day 29 or Day 113: number analyzed (Participants) | 83 | 94 | 42 | 45
  Against WCE: Either Day 29 or Day 113 | 54 | 64 | 21 | 11
  Against PT, FHA, PRN: Either Day 29 or Day 113: number analyzed (Participants) | 83 | 94 | 41 | 45
  Against PT, FHA, PRN: Either Day 29 or Day 113 | 23 | 14 | 5 | 2
  Against at least 2 of WCE, PT, FHA, or PRN: Any of Days 29, 78, or 113: number analyzed (Participants) | 83 | 94 | 42 | 45
  Against at least 2 of WCE, PT, FHA, or PRN: Any of Days 29, 78, or 113 | 64 | 70 | 23 | 11
  Against at least 2 of WCE, PT, FHA, or PRN: Either Day 169 or Day 254: number analyzed (Participants) | 75 | 90 | 37 | 39
  Against at least 2 of WCE, PT, FHA, or PRN: Either Day 169 or Day 254 | 47 | 43 | 17 | 3
  Boosting achieved on Day 113 (over Day 78) against WCE: number analyzed (Participants) | 77 | 89 | 38 | 40
  Boosting achieved on Day 113 (over Day 78) against WCE | 23 | 7 | 11 | 6

11. Secondary Outcome: Mucosal Immunogenicity - Summary of GMFRs of Mucosal Absolute S-IgA/Total S-IgA Against Whole Cell Extract by Vaccine Group and Time Point
Description: Mucosal Immunogenicity: Summary of GMFRs of Mucosal Absolute S-IgA/Total S-IgA Against Whole Cell Extract by Vaccine Group and Time Point - GMFRs on Day 29 and Day 78 over baseline (Day 1)
Time Frame: Days 29 and 78
Population: 10^9 Immunogenicity Analysis Set. The Day 29 and Day 78 GMFR values are for the pooled BPZE1 group (BPZE1/BPZE1 + BPZE1/placebo) and pooled Boostrix group (Boostrix/BPZE1 + Boostrix/placebo), since these Days are prior to the Day 85 challenge/boost. The number analyzed includes participants with nonmissing values.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | BPZE1 Intranasal Prime, BPZE1 Boost | Boostrix IM Prime, BPZE1 Boost
Number analyzed (Participants) | 179 | 88
Ratio
  GMFR WCE Day 29: number analyzed (Participants) | 173 | 87
  GMFR WCE Day 29 | 2.22 [1.94 to 2.54] | 1.07 [0.92 to 1.24]
  GMFR WCE Day 78: number analyzed (Participants) | 174 | 82
  GMFR WCE Day 78 | 2.10 [1.84 to 2.39] | 1.04 [0.89 to 1.22]

12. Secondary Outcome: Mucosal Immunogenicity - Summary of GMFRs of Mucosal Absolute S-IgA/Total S-IgA Against Whole Cell Extract by Vaccine Group and Time Point
Description: Mucosal Immunogenicity: Summary of GMFRs of Mucosal Absolute S-IgA/Total S-IgA Against Whole Cell Extract by Vaccine Group and Time Point - GMFRs on Day 113, Day 169, and Day 254 over baseline (Day 1)
Time Frame: Days 113, 169, 254
Population: 10^9 Immunogenicity Analysis Set. Note: Participants who were randomized to receive BPZE1 as the second vaccination (ie, revaccination/attenuated challenge) but who did not receive a second vaccination and continued in the study after second vaccination were placed into the BPZE1/Placebo or Boostrix/Placebo group according to first vaccine received. The number analyzed includes participants with nonmissing values.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | BPZE1 Intranasal Prime, BPZE1 Boost | BPZE1 Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 Boost | Boostrix IM Prime, Placebo Boost
Number analyzed (Participants) | 85 | 94 | 43 | 45
Ratio
  GMFR WCE Day 113: number analyzed (Participants) | 75 | 89 | 38 | 40
  GMFR WCE Day 113 | 2.96 [2.35 to 3.75] | 2.04 [1.71 to 2.43] | 1.91 [1.53 to 2.37] | 1.15 [0.94 to 1.39]
  GMFR WCE Day 169: number analyzed (Participants) | 75 | 88 | 35 | 39
  GMFR WCE Day 169 | 2.23 [1.80 to 2.77] | 1.57 [1.33 to 1.86] | 1.75 [1.39 to 2.19] | 0.82 [0.67 to 0.99]
  GMFR WCE Day 254: number analyzed (Participants) | 71 | 86 | 36 | 37
  GMFR WCE Day 254 | 1.73 [1.39 to 2.15] | 1.45 [1.22 to 1.72] | 1.26 [1.02 to 1.55] | 0.82 [0.68 to 0.99]

13. Secondary Outcome: Colonization - Summary of Colonization for B. Pertussis Bacterial Culture From Nasal Sample by Timepoint
Description: Number of participants with positive B. pertussis by bacterial culture of nasal sample on any of Days 92, 96, and 113 (colonization)
Time Frame: Days 92, 96, 113
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 Intranasal Prime, BPZE1 Boost | BPZE1 Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 Boost | Boostrix IM Prime, Placebo Boost
Number analyzed (Participants) | 80 | 91 | 40 | 41
Participants | 8 | 0 | 28 | 0

14. Secondary Outcome: Safety - Number of Participants With Unsolicited AEs
Description: Number of participants with Unsolicited AEs collected Day 1 to Day 29 by Medical Dictionary for Regulatory Activities (MedDRA) classification.
  Threshold is greater than or equal to 5% of participants.
Time Frame: Days 1 through 29
Population: 10^9 Safety Analysis Set. Note: Participants who were randomized to receive BPZE1 as the second vaccination (ie, revaccination/attenuated challenge) but who did not receive a second vaccination and continued in the study after second vaccination were placed into the BPZE1/Placebo or Boostrix/Placebo group according to first vaccine received.
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 Intranasal Prime, BPZE1 Boost | BPZE1 Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 Boost | Boostrix IM Prime, Placebo Boost
Number analyzed (Participants) | 87 | 96 | 46 | 50
Participants
  Headache | 5 | 7 | 0 | 1
  Nasal congestion | 5 | 4 | 3 | 3
  Rhinorrhoea | 5 | 3 | 2 | 2
  Sneezing | 6 | 2 | 2 | 1

15. Secondary Outcome: Safety - Number of Participants With Unsolicited AEs
Description: Number of participants with Unsolicited AEs Day 85 through Day 113 by MedDRA classification.
  Threshold is greater than or equal to 5% of participants.
Time Frame: Days 85 through 113
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 Intranasal Prime, BPZE1 Boost | BPZE1 Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 Boost | Boostrix IM Prime, Placebo Boost
Number analyzed (Participants) | 87 | 96 | 46 | 50
Participants
  Upper respiratory tract infection | 4 | 5 | 0 | 4
  Nasal congestion | 1 | 6 | 4 | 4

16. Secondary Outcome: Safety - Number of Participants With Serious AEs
Description: Number of participants with Serious AEs collected on Day 1 through Day 84 by MedDRA classification.
Time Frame: Days 1 to 84
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 Intranasal Prime, BPZE1 Boost | BPZE1 Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 Boost | Boostrix IM Prime, Placebo Boost
Number analyzed (Participants) | 87 | 96 | 46 | 50
Participants
  Bacterial sepsis | 0 | 1 | 0 | 0
  Cellulitis | 0 | 1 | 0 | 0
  Post procedural haemorrhage | 1 | 0 | 0 | 0
  Hyperglycaemia | 0 | 1 | 0 | 0

17. Secondary Outcome: Safety - Number of Participants With Serious AEs
Description: Number of participants with Serious AEs collected on Day 85 through Day 113 by MedDRA classification.
Time Frame: Days 85 to 113
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 Intranasal Prime, BPZE1 Boost | BPZE1 Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 Boost | Boostrix IM Prime, Placebo Boost
Number analyzed (Participants) | 87 | 96 | 46 | 50
Participants
  Diabetic metabolic decompensation | 0 | 1 | 0 | 0
  Other | 0 | 0 | 0 | 0

18. Secondary Outcome: Safety - Number of Participants With Serious AEs
Description: Number of participants with Serious AEs collected on Day 114 through Day 254 by MedDRA classification.
Time Frame: Days 114 to 254 (end of study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 Intranasal Prime, BPZE1 Boost | BPZE1 Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 Boost | Boostrix IM Prime, Placebo Boost
Number analyzed (Participants) | 87 | 96 | 46 | 50
Participants
  Obesity | 0 | 0 | 1 | 0
  Other | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Unsolicited treatment-emergent adverse events (TEAEs) - Days 1 through 29 and Days 85 through 113; All-cause mortality and SAEs - Days 1 through 254 (end of study)
Description: 10^7 and 10^9 Safety Analysis Set (includes 10^9 Safety Analysis Set [n=279] and Safety Lead-in Cohort of participants who received BPZE1 10^7 CFU [n=20]). Participants who were randomized to receive BPZE1 as the second vaccination (ie, revaccination/attenuated challenge) but who did not receive a second vaccination and continued in the study after second vaccination were placed into the BPZE1/Placebo or Boostrix/Placebo group according to first vaccine received.
Groups:
- BPZE1 Intranasal Prime, BPZE1 Boost: Individual will receive an intranasal dose of BPZE1 via the VaxINator atomization device and a dose of IM placebo on Day 1. Individuals will receive a boost dose of intranasal BPZE1 via the VaxINator™ atomization device on Day85. (10^9 Safety Analysis Set)
- BPZE1 Intranasal Prime, Placebo Boost: Individual will receive an intranasal dose of BPZE1 via the VaxINator atomization device and a dose of IM placebo on Day 1. Individuals will receive a boost dose of intranasal placebo via the VaxINator™ atomization device on Day 85. (10^9 Safety Analysis Set)
- Boostrix IM Prime, BPZE1 Boost: Individual will receive an intranasal dose of placebo via the VaxINator atomization device and a dose of IM Boostrix (aP vaccine comparator) on Day 1. Individuals will receive a boost dose of intranasal BPZE1 via the VaxINator™ atomization device on Day 85. (10^9 Safety Analysis Set)
- Boostrix IM Prime, Placebo Boost: Individual will receive an intranasal dose of placebo via the VaxINator atomization device and a dose of IM Boostrix (aP vaccine comparator) on Day 1. Individuals will receive a boost dose of intranasal placebo via the VaxINator™ atomization device on Day 85. (10^9 Safety Analysis Set)
Arm/Group | BPZE1 Intranasal Prime, BPZE1 Boost | BPZE1 Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 Boost | Boostrix IM Prime, Placebo Boost | BPZE1 (10^7) Intranasal Prime, BPZE1 (10^7) Boost | BPZE1 (10^7) Intranasal Prime, Placebo Boost | Boostrix IM Prime, BPZE1 (10^7) Boost
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/96 | 0/46 | 0/50 | 0/8 | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/87 | 3/96 | 1/46 | 0/50 | 0/8 | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 25/87 | 26/96 | 14/46 | 12/50 | 3/8 | 2/8 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BPZE1 Intranasal Prime, BPZE1 Boost (N=87) | BPZE1 Intranasal Prime, Placebo Boost (N=96) | Boostrix IM Prime, BPZE1 Boost (N=46) | Boostrix IM Prime, Placebo Boost (N=50) | BPZE1 (10^7) Intranasal Prime, BPZE1 (10^7) Boost (N=8) | BPZE1 (10^7) Intranasal Prime, Placebo Boost (N=8) | Boostrix IM Prime, BPZE1 (10^7) Boost (N=4)
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BPZE1 Intranasal Prime, BPZE1 Boost (N=87) | BPZE1 Intranasal Prime, Placebo Boost (N=96) | Boostrix IM Prime, BPZE1 Boost (N=46) | Boostrix IM Prime, Placebo Boost (N=50) | BPZE1 (10^7) Intranasal Prime, BPZE1 (10^7) Boost (N=8) | BPZE1 (10^7) Intranasal Prime, Placebo Boost (N=8) | Boostrix IM Prime, BPZE1 (10^7) Boost (N=4)
Headache (Nervous system disorders) | 5 | 7 | 0 | 1 | 0 | 0 | 0 — Days 1-29
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 3 | 3 | 0 | 0 | 0 — Days 1-29
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 2 | 2 | 0 | 0 | 0 — Days 1-29
Sneezing (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 2 | 1 | 0 | 0 | 0 — Days 1-29
Upper respiratory tract infection (Infections and infestations) | 4 | 5 | 1 | 4 | 0 | 0 | 0 — Days 85-113
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 4 | 4 | 1 | 0 | 0 — Days 85-113
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Days 1-29
Coagulation test abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Days 1-29
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 — Days 1-29
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 — Days 1-29
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0 — Days 1-29
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Days 1-29
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Days 1-29
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 — Days 1-29
Malaise (General disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 — Days 85-113
Burns first degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Days 85-113
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Days 85-113
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 — Days 85-113
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 — Days 85-113

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Protocol Section 10.9: After study completion, data may be considered for reporting at scientific meeting/publication in scientific journal. In these cases, sponsor will be responsible for these activities to determine how the manuscript is written/edited, number/order of authors, publication for submission, etc. Sponsor has final approval over all issues.

Data are property of sponsor and cannot be published without prior authorization, but data/publication thereof will not be unduly withheld.

DOCUMENTS (2):
  • Study Protocol (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT03942406/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT03942406/SAP_001.pdf